CLINICAL TRIAL: NCT07093528
Title: CMR Substudy of Coronary Sinus Reducer for the Management of Symptomatic Heart Failure With a Preserved Ejection Fraction (HFpEF) Associated With Coronary Microvascular Dysfunction (CMD)
Brief Title: A Study Of CS Reducer For Symptomatic Heart Failure With HFpEF And CMD
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Claire E. Raphael, Principal Investigator, Mayo Clinic
Other Study IDs: 25-005812
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Coronary Microvascular Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Failure with a Preserved Ejection Fraction (HFpEF): Subjects with diagnosed Heart failure with a preserved ejection fraction (HFpEF), non-obstructive Coronary Artery Disease (CAD), and have documented CMD.
  Interventions: Diagnostic Test: Cardiovascular Magnetic Resonance (CMR)

INTERVENTIONS:
Diagnostic Test: Cardiovascular Magnetic Resonance (CMR) — Patients will consent to undergo a 50-minute non-invasive stress perfusion CMR.

SUMMARY:
To evaluate the effect of CS reducer implantation in patients with HFPEF and CMD on myocardial ischemia, measured by stress myocardial perfusion using cardiovascular magnetic resonance (CMR)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Enrollment in main CS-reducer HFPEF study IRB# 25-002292

Exclusion Criteria:

* Metal implants that are not suitable for MRI
* Inability or unwillingness of individual to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects included in the main CS-reducer HFPEF study (IRB# 25-002292)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in endocardial:epicardial perfusion ratio | Baseline, 6 Months
  Endocardial:Epicardial Perfusion Ratio is a measure of myocardial blood flow and will be determined by Cardiovascular magnetic resonance (CMR)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Raphael, M.B.B.S., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No